CLINICAL TRIAL: NCT04048902
Title: Effects of Shortwave Diathermy and Pilates Exercises in Patients With Chronic Non-specific Low Back Pain: a Protocol of a Randomized Controlled Trial
Brief Title: Shortwave Diathermy and Pilates Exercises in Patients With Chronic Non-specific Low Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Raquel A. Casarotto, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48391615.9.0000.0065
Record Dates: First submitted 2019-04-15; First posted 2019-08-07 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain
Keywords: Exercise Therapy; Clinical Trial; Diathermy; Physical Therapy Modalities
MeSH Terms: conditions — Low Back Pain; Fever

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates and Shortwave placebo (Placebo Comparator): In this group the patients will receive 20 minutes of short wave placebo application. The equipment will keep the timer on and the intensity will remain at zero. The patient will be informed that the dose is subsensory and therefore there will be no perception of the passage of the short waves through the body.The application will be performed with two coplanar plates in parallel, arranged on the right and left side of the lumbar region, maintaining a distance of 5 to 10 cm between them, with the patient lying in the dorsal decubitus position
  Interventions: Device: Pilates and Shortwave placebo
- Pilates and Shortwave active (Active Comparator): In this group the patients will receive 20 minutes of application of the Shortwave Active continuous mode (thermal effect), with vigorous local thermal sensation.The application will be performed with two coplanar plates in parallel, arranged on the right and left side of the lumbar region, maintaining a distance of 5 to 10 cm between them, with the patient lying in the dorsal decubitus position
  Interventions: Device: Pilates and Shortwave active

INTERVENTIONS:
Device: Pilates and Shortwave placebo — Pilates exercises and application of the device without produce thermal effects
  Arms: Pilates and Shortwave placebo
Device: Pilates and Shortwave active — Pilates exercises and application of the device producing thermal effects
  Arms: Pilates and Shortwave active

SUMMARY:
The aim of this study is to verify the effectiveness of the association of Shortwave Diathermy and Pilates exercises in patients with chronic non-specific low back pain, on the reduction of pain, functional disability and improvement of the quality of life.

DETAILED DESCRIPTION:
The drawing of the study will be a prospective, randomized controlled trial and double-blind with quantitative approach. Study participants 36 subjects diagnosed with non-specific chronic low back pain, which will be divided in two groups with 18 subjects in each: experimental group, which will be submitted to placebo + exercise shortwave diathermy and the control group to do active + exercise shortwave diathermy. There will be 12 one-hour sessions twice a week. The subjects will apply Shortwave Diathermy for 20 minutes, followed by Pilates mat.

ELIGIBILITY:
Inclusion Criteria:

* individuals diagnosed with chronic non-specific low back pain for a period of more than 3 months, without irradiation for lower limbs;
* who present pain intensity greater than 3 points in the Numerical Pain Scale;
* to sign the Free and Informed Consent Form.

Exclusion Criteria:

* BMI> 30;
* previous surgeries in the spine;
* severe spinal affection (tumors, infection, unconsolidated or vicious consolidation fractures, inflammatory diseases);
* rheumatic disease;
* contraindication to performing the exercises according to the American College of Sports Medicine Guidelines;
* degenerative or inflammatory joint and other body segments;
* patients who are in labor litigation;
* pregnancy;
* patients who are undergoing other type of physiotherapeutic or drug treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in pain through Pain visual analogue scale | Before the treatment, up to 3, 6 and 18 weeks
  Scale with 11 centimeters is used for evaluate pain intensity, being "0" no pain and "10" the worst possible pain
Change in pain through The McGill pain questionnaire | Before the treatment, up to 3, 6 and 18 weeks
  It is organized in four categories: sensory, affective, evaluative and mixed, with 20 subcategories and 78 words descriptors of pain, describing the quality of pain. The pain evaluation index is the sum of the values added, and each word chosen in each dimension is the maximum score of each category: Sensory = 34, Affective = 17, Evaluative = 5, Mixed = 11, Total = 67.

SECONDARY OUTCOMES:
Functional disability | Before the treatment, up to 3, 6 and 18 weeks
  The Rolland and Morris Questionnaire, validated in Brazil, will quantify the functional limitations caused by low back pain. The questionnaire is composed of 24 questions related to normal activities of daily living, in which each affirmative answer corresponds to a point. The final score is determined by the sum of the values obtained. Values close to zero represent the best results (lower limitation), and values close to 24 the worst results. Values above 14 points are considered as a severe spinal impairment.
Patients' perceptions of their health-related quality of life: The Short-Form Health Survey questionnaire (SF-36) | Before the treatment, up to 3, 6 and 18 weeks
  The Short-Form Health Survey questionnaire (SF-36) will assess the health-related quality of life of patients. This instrument contains 36 questions grouped into eight areas: functional capacity (10 items), physical aspects (2 items), pain (2 items), general state of health (5 items), vitality (4 items), social aspects (2 items), emotional (3 items) and mental health (5 items). The values in each domain vary from 0 to 100 and, more indicate a better quality of life.
Perception of global effect | Before the treatment, up to 3, 6 and 18 weeks
  Evaluates the level of perception of patient recovery through a Scale Numbers of 11 points comparing the onset of symptoms at the beginning of treatment in relation to the last days. It varies from -5 to +5, being -5: extremely worse; zero: no modification; and +5: fully recovered, with the highest score representing greater recovery.
Emotional Functioning | Before the treatment, up to 3, 6 and 18 weeks
  It will be evaluated by the Brazilian version of the Visual Analog Scale for anxiety. Analogic visual scale for anxiety is a horizontal line of 100 mm in length. The tip left without anxiety and the right tip means worse anxiety.
Depressive Symptom | Before the treatment, up to 3, 6 and 18 weeks
  It will be evaluated by the Brazilian version of the Beck Depression Inventory, a self-assessment measure of depression. It is a questionnaire with 21 items whose intensity ranges from 0 to 3 points. Largest scores indicate more depressive symptoms.
Symptoms and adverse events | Before the treatment, up to 3, 6 and 18 weeks
  The record of the symptoms and adverse events that occurred during the established behavior will be captured passively through spontaneous reports of the patient. The active catch will use a questionnaire with a record of the duration and intensity of the adverse symptom reported by the patient. You will then be asked to the patient graduates the certainty of their affirmations according to a Likert scale (being 1 not certain and 5 total certainty).
Patient Satisfaction: The MedRisk scale | Patients will be evaluated up to 6 weeks
  The MedRisk scale consists of 20 items, 10 items related to the therapist-patient interaction; 8 items involving evaluation of the infrastructure and work organization of the physical therapy clinic and 2 items that are considered as global evaluation of the treatment. The patient elects level of satisfaction in each item by selecting a Likert scale ranging from 1 "completely disagree" to 5 "agree completely" or through an option "not applicable", with high scores representing high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel A Casarotto, PhD, Principal Investigator — University of Sao Paulo; Sandra Amaral, Bachelor, Principal Investigator — University of Sao Paulo
Locations (1):
- Department of Physical Therapy, Speech and Occupational Therapy of University of São Paulo, São Paulo, Brazil